CLINICAL TRIAL: NCT05083442
Title: A Feasibility Study Addressing the Adjunct Use of Low-Level Laser to Mayo Lifestyle Modification Education and Wellness Coaching for Reducing Central Adiposity and Fat Mass
Brief Title: Low-level Laser and Lifestyle Modifications
Acronym: LLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Erchonia Corporation (Industry)
Responsible Party: Principal Investigator, Ivana T Croghan, PhD, Professor of Medicine, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-008379
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Overweight and Obesity; Weight Loss
Keywords: BMI; Fat Mass; Weight Loss; Body Circumference Reduction
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Low-Level Light Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial where subjects are placed into 2 different study arms. Subjects randomized to 2 groups that either receive Low Level Laser therapy with lifestyle modifications or Sham (placebo) with Lifestyle Modifications.
Who Masked: Participant
Masking Description: Randomization will be set up by a statistician through REDCap, the data collection system utilized for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 - LLLT (Active Comparator): Subject receive Laser treatments and Lifestyle Modifications
  Interventions: Device: Low Level Laser Therapy
- Group 2 - SHAM (Sham Comparator): Subject receives Sham Laser treatments and Lifestyle Modifications
  Interventions: Other: Sham (placebo)

INTERVENTIONS:
Device: Low Level Laser Therapy — Non-surgical cosmetic treatment which can be used by individuals intending to reduce size of the mid-section
  Arms: Group 1 - LLLT
Other: Sham (placebo) — Use of sham (placebo) option
  Arms: Group 2 - SHAM

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of Low Level Laser Therapy in combination with Lifestyle Modifications in helping people reduce the extra weight and size in the central body region

DETAILED DESCRIPTION:
Subjects will undergo Low Level Laser Therapy or Sham (placebo) treatments while incorporating lifestyle modifications through of wellness coaching.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. have a BMI 25-39.9 kg/m2
3. be able to participate fully in all aspects of the study; and
4. have understood and signed study informed consent

Exclusion Criteria:

1. have used weight loss medications or participated in a weight loss program within the past 30 days
2. are currently taking medications or supplements known to affect weight, such as insulin or sulfonylurea, prednisone or garcinia cambrogia
3. have had weight fluctuations of 5 pounds or more in the past month
4. have an implanted device (including pacemaker or lap band) in the targeted area of LLLT
5. have a known active eating disorder
6. have a known, active, untreated clinically significant psychiatric condition (alcohol or substance abuse, psychosis, bipolar disorder, or depression)
7. have used an investigational drug within 30 days of study enrollment
8. Reports being currently pregnant, lactating, or are of child-bearing potential or are likely to become pregnant during the low-level laser therapy treatment phase and are unwilling to use a reliable form of contraception. Acceptable forms include:

   1. Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
   2. Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
   3. Intrauterine device (IUD)
   4. Total hysterectomy or tubal ligation
   5. Abstinence (no sex)
9. have a history of any major cardiovascular events including heart valve disease, ongoing angina, cardiac arrhythmias, congestive heart failure, acute coronary syndrome, stroke, transient ischemic attack, or peripheral vascular disease
10. have current uncontrolled hypertension (systolic > 160 mm Hg or diastolic > 95 mm Hg) documented on 2 separate occasions
11. have clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, lymphatic, respiratory, or metabolic disease (such as uncontrolled diabetes type 2) or active cancer or are within 1 year of cancer remission
12. surgical intervention for body sculpting/weight loss, such as liposuction, abdominoplasty, stomach stapling, lap band surgery, etc. within 12 months prior to enrollment
13. medical, physical, or other contraindications for body sculpting/weight loss
14. any medical condition known to affect weight levels and/or to cause bloating or swelling
15. a diagnosis of, and/or taking medication for, irritable bowel syndrome
16. active infection, wound or other external trauma to the areas to be treated with the laser
17. known photosensitivity disorder
18. current active cancer or currently receiving treatment for cancer; or
19. have a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana T Croghan, PhD, Principal Investigator — Professor of Medicine, College of Medicine; Ryan T Hurt, MD, PhD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited from the local community through internet postings, Mayo Clinic physician referrals, and word of mouth.
Period: Overall Study
Arm/Group | Group 1 - LLLT | Group 2 - SHAM
Started | 30 | 30
Completed | 27 | 24
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — scheduling difficulties | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - LLLT | Group 2 - SHAM | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (10.1) | 37.7 (11.7) | 39.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 3 | 8 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race/ethnicity: white, not hispanic | 28 | 26 | 54
  race/ethnicity: other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat Mass From Baseline to 6 Weeks
Description: The change in fat mass from baseline to the end of treatments at 6 weeks
Time Frame: 6 weeks
Population: Analysis population includes subjects with non-missing values for given outcome (change in fat mass at 6 weeks)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Group 1 - LLLT | Group 2 - SHAM
Number analyzed (Participants) | 25 | 24
Kg | -1.3 (1.5) | -2.0 (2.4)
Statistical Analysis 1: Comparison: Group 1 - LLLT vs Group 2 - SHAM; Groups were compared using analysis of covariance with baseline included as the covariate; Test type: Superiority; p = 0.19, ANCOVA; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.4 to 1.9] — Estimated difference between groups from analysis of covariance with baseline fat mass included as the covariate

2. Primary Outcome: Change in Waist Circumference From Baseline to 6 Weeks
Description: The change in waist circumference from baseline to the end of treatments at 6 weeks
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group 1 - LLLT | Group 2 - SHAM
Number analyzed (Participants) | 25 | 24
cm | -1.8 (3.5) | -1.8 (4.0)
Statistical Analysis 1: Comparison: Group 1 - LLLT vs Group 2 - SHAM; Groups were compared using analysis of covariance with baseline included as the covariate; Test type: Superiority; p = 0.745, ANCOVA; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.5 to 2.1] — Estimated difference between groups from analysis of covariance with baseline fat mass included as the covariate

ADVERSE EVENTS:
Time Frame: AE's were collected over the 6 weeks of the LLLT intervention.
Arm/Group | Group 1 - LLLT | Group 2 - SHAM
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 6/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - LLLT (N=30) | Group 2 - SHAM (N=30)
Loose Stool (Gastrointestinal disorders) | 3 (3) | 0 (0)
muscle contraction/tingling (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
stomach/gas pain (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT05083442/Prot_SAP_000.pdf